CLINICAL TRIAL: NCT03035799
Title: A Randomized Trial Comparing Two Types of Diets on Psychological and Gastrointestinal Symptoms
Brief Title: Comparing Two Types of Diets on Psychological and Gastrointestinal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00082222
Record Dates: First submitted 2017-01-18; First posted 2017-01-30 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Paleolithic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paleolithic Diet (Experimental): Paleolithic Diet
  Interventions: Other: Paleolithic diet
- General Healthful Diet (Active Comparator): General Healthful Diet
  Interventions: Other: General Healthful Diet

INTERVENTIONS:
Other: Paleolithic diet — Paleolithic diet
  Arms: Paleolithic Diet
Other: General Healthful Diet — General Healthful Diet
  Arms: General Healthful Diet

SUMMARY:
This pilot study proposes to gain a better understanding of the health benefits of the popular "paleo-diet" in patients with irritable bowel syndrome (IBS) and explore underlying mechanisms of benefit.

DETAILED DESCRIPTION:
In the proposed study, the primary hypothesis is that, compared with a customary diet, consumption of a paleo-diet will improve psychological and gastrointestinal symptoms in patients with irritable bowel syndrome. Investigators also hypothesize consumption of the Paleolithic diet will result in decreased intestinal permeability, decreased inflammatory markers, and changes in the gut microbiome and microbiologic profiles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate Irritable Bowel Syndrome (IBS) and mild to moderate anxiety or depression
* Other causes of bowel symptoms excluded to the satisfaction of the Study Team
* Age at least 18 years at initial screening visit
* Patients who are able to sign and understand the study's informed consent form
* Patients able to complete all screening evaluations and procedures

Exclusion Criteria:

* Patients in inpatient hospital care
* Severe or refractory bowel or psychological symptoms
* Current consumption of a Paleolithic diet
* Known Celiac disease
* Uncontrolled thyroid disease as indicated by an abnormal thyroid stimulating hormone (TSH) level
* Uncontrolled diabetes as indicated by a HbA1c equal to 6.5 or greater
* Patients unable to speak English
* Inability to obtain informed consent
* Pregnant or nursing women
* Any condition, which in the opinion of the investigator, would interfere with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Vitality | The change between baseline and 4 weeks (post-intervention).
  Vitality as measured on the vitality subscale of the short form health survey (SF36). This instrument assesses vitality (energy level and fatigue) and is a subscale of SF36, a general health survey designed for use in clinical practice and research, health policy evaluation and general population surveys. The Vitality Subscale score is determined by responses to 4 items: Did you feel full of life? Did you have a lot of energy? Did you feel worn out? Did you feel tired? The lower the score the more disability. The higher the score the less disability.

SECONDARY OUTCOMES:
Anxiety | The change between baseline and 4 weeks (post-intervention).
  Anxiety as measured by the Generalized Anxiety Disorder 7-item (GAD-7) questionnaire.
  GAD-7 Questionnaire: This is a 7 item inventory rated on a 4 point Likert-type scale. Its purpose is to allow for brief and accurate detection of anxiety as well as for longitudinal anxiety symptom evaluation. Lower scores indicate less severe symptoms and higher scores equal more severe symptoms.
Depression | The change between baseline and 4 weeks (post-intervention).
  Depression as measured by the Patient Health Questionnaire-9' (PHQ-9) questionnaire.
  PHQ-9: This is a 9 item inventory rated on a 4 point Likert-type scale. Its purpose is to allow for brief and accurate diagnosis of depression as well as for longitudinal depression symptom evaluation. Lower scores indicate less severe symptoms and higher scores equal more severe symptoms.
Activity level | The change between baseline and 4 weeks (post-intervention).
  Activity level/amount of exercise as measured by the Godin Leisure-Time Exercise Questionnaire. The Godin Leisure-Time Exercise Questionnaire is a simple questionnaire to measure a person's leisure time exercise. It is designed to be reliable valid and easy to complete quickly without a need for detailed review. Lower scores indicate less activity and higher scores equal more activity.
Gastrointestinal symptoms | The change between baseline and 4 weeks (post-intervention).
  Gastrointestinal symptoms as measured by the NIH-Promis Gastrointestinal Symptom Scale
  a. NIH-Promis Gastrointestinal Symptom Scales for 8 domains: Gastroesophageal reflux (13 items), disrupted swallowing (7 items), diarrhea (5 items), bowel incontinence/soilage (4 items), nausea and vomiting (4 items), constipation (9 items), belly pain (6 items), and gas/bloat/flatulence (12 items). Lower scores indicate less severe symptoms and higher scores equal more severe symptoms.
Visceral sensitivity | The change between baseline and 4 weeks (post-intervention).
  Visceral sensitivity as measured by the Visceral Sensitivity Index. Visceral Sensitivity Index assesses gastrointestinal-specific anxiety, the cognitive, affective, and behavioral response to fear of gastrointestinal sensations, symptoms, and the context in which these visceral sensations and symptoms occur. Lower scores indicate less severe symptoms and higher scores equal more severe symptoms.
Overall health status (Short Health Scale) | The change between baseline and 4 weeks (post-intervention).
  Overall health status as measured by the Short Health Scale questionnaires. The "Short Health Scale" is a 4-item questionnaire covering aspects of subjective health. Lower scores indicate less severe symptoms and higher scores equal more severe symptoms.
Overall health status (EQ-5D) | The change between baseline and 4 weeks (post-intervention).
  Overall health status (global health outcomes measure) as measured by the EuroQol 5 Dimension (EQ-5D) The EQ-5D descriptive system consists of five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. Scores range from 5-25, with higher scores indicating more severe symptoms/decreased quality of life.descriptive system consists of five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. Lower scores indicate less severe symptoms and higher scores equal more severe symptoms.

OTHER OUTCOMES:
Intestinal permeability | The change between baseline and 4 weeks (post-intervention).
  Change in intestinal permeability as measured by plasma zonulin levels
Change in inflammatory markers | The change between baseline and 4 weeks (post-intervention).
  Change in inflammatory markers as measured by serum C-reactive protein levels
Change in stool metabolomics | The change between baseline and 4 weeks (post-intervention).
  Change in stool metabolomics as measured by stool metabolite testing.
Change in stool microbiome profile | The change between baseline and 4 weeks (post-intervention).
  Change in stool microbiota profile as measured by 16S DNA sequencing of stool samples.
Biobank specimen collection of urine. | The change between baseline and 4 weeks (post-intervention).
  Biobank specimen collection of stool, blood, urine, and saliva to be studied in future studies
Biobank specimen collection of stool. | The change between baseline and 4 weeks (post-intervention).
  Biobank specimen collection of stool, blood, urine, and saliva to be studied in future studies
Biobank specimen collection of saliva. | The change between baseline and 4 weeks (post-intervention).
  Biobank specimen collection of stool, blood, urine, and saliva to be studied in future studies
Biobank specimen collection of blood. | The change between baseline and 4 weeks (post-intervention).
  Biobank specimen collection of stool, blood, urine, and saliva to be studied in future studies

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Pasricha, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided